CLINICAL TRIAL: NCT02499653
Title: A Psychological Intervention to Promote Acceptance and Adherence to Non-Invasive Ventilation (NIV) in People With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: A Psychological Intervention to Promote Acceptance and Adherence to NIV in People With COPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Collaborators: Catholic University of the Sacred Heart (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FDG_PSYNIV_COPD01
Record Dates: First submitted 2015-06-29; First posted 2015-07-16 (Estimated); Last update posted 2018-02-06 (Actual); Status verified 2016-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Chronic Obstructive Pulmonary Disease (COPD); Non Invasive Ventilation (NIV); Acceptance; Adherence; Clinical Psychology
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Psychosocial Intervention; Videotape Recording

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Psychological Intervention (Experimental): In addition to the standard care, subjects are participating in a brief psychological support, which will include elements of psychological well-being's promotion and cognitive restructuring exercises (mindfulness).
  Interventions: Behavioral: Psychological Intervention
- Videos (Active Comparator): The subjects assigned in the Control Group watch some videos relating to the management of their disease.
  Interventions: Behavioral: Videos

INTERVENTIONS:
Behavioral: Psychological Intervention
  Arms: Psychological Intervention
Behavioral: Videos
  Arms: Videos

SUMMARY:
This study aims to analyze the impact of a brief psychological support intervention in the promotion of the adherence to Non Invasive Ventilation (NIV) among people with Chronic Obstructive Pulmonary Disease (COPD). The investigators expect to see a positive impact of this intervention on both physical and psychological well-being, and consequently, a reduction of health costs.

ELIGIBILITY:
Inclusion Criteria:

* age> or =18 years
* the voluntary participation to the Study
* inpatients or outpatients
* subjects with Chronic Obstructive Pulmonary Disease (COPD), from moderate (GOLD 2- 50% ≤ FEV1 <80% pred.) to severe (GOLD 3- 30% ≤ FEV1 <50%pred.) (FEV1= Forced Expiratory Volume in the 1st Second)

Exclusion Criteria:

* refusal of the Informant Consent
* pregnancy
* subjects affected by oncological or psychiatric illnesses
* immune depressive condition as the principal condition
* usage of antidepressant drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2015-06; Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Quality of Life (QoL) in COPD patients at 3, 6 and 12 months as measured by EuroQoL (EQ5D) | Baseline + After 3, 6 and 12 months following the recruitment
  EuroQoL or EQ5D, a simple and short questionnaire consists of two distinct sections: the first in which there are five items (mobility, self-care, usual activities, pain / discomfort, anxiety / depression), concerning the status of health of the subject, which is required to indicate the severity level; the second section includes a visual-analogue scale instead represented graphically as a thermometer graduated from 0 (worst possible health status) to 100 (best possible health state), on which the respondent must indicate the level of perceived health at the time. All subjects will be assigned to psychometric assessment.

SECONDARY OUTCOMES:
Change from baseline in acceptance NIV in COPD patients at 3, 6 and 12 months as measured by weekly means and standard deviations of hours of use of Non Invasive Ventilation (NIV) | Baseline + After 3, 6 and 12 months following the recruitment
  It will be summarized by weekly means and standard deviations of hours of use of Non Invasive Ventilation (NIV). All subjects will be assigned to this assessment.
Change from baseline in adherence NIV in COPD patients at 3, 6 and 12 months as measured by a modified version of the Beliefs About Medicine Questionnaire (BMQ) | Baseline + After 3, 6 and 12 months following the recruitment
  A specific instrument, adapted to detect representations of NIV, it is being validated. It will be based on a modified version of the Beliefs about Medicines Questionnaire (BMQ) developed by Prof. Dr. Rob Horne et al. This tool is used to check the patient's beliefs regarding medications. It consists of two scales: Beliefs Specifications (10 items) and General Beliefs (8 items). In order to achieve the objectives of the study, we will use a modified version of the BMQ, adapted to detect representations of NIV. The unit of measure will be the scale that emerges from the test. All subjects will be assigned to psychometric assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- Paolo Banfi, Milan, Italy

REFERENCES:
- [Background] Balestroni G, Bertolotti G. [EuroQol-5D (EQ-5D): an instrument for measuring quality of life]. Monaldi Arch Chest Dis. 2012 Sep;78(3):155-9. doi: 10.4081/monaldi.2012.121. Italian. PMID 23614330
- [Result] Horne, R., Weinman, J., & Hankins, M. (1999). The beliefs about medicines questionnaire: the development and evaluation of a new method for assessing the cognitive representation of medication. Psychology and health, 14(1), 1-24.
- [Derived] Volpato E, Banfi P, Pagnini F. Promoting Acceptance and Adherence to Noninvasive Ventilation in Chronic Obstructive Pulmonary Disease: A Randomized Controlled Trial. Psychosom Med. 2022 May 1;84(4):488-504. doi: 10.1097/PSY.0000000000001053. Epub 2022 Feb 10. PMID 35149638
- [Derived] Volpato E, Banfi P, Pagnini F. A psychological intervention to promote acceptance and adherence to non-invasive ventilation in people with chronic obstructive pulmonary disease: study protocol of a randomised controlled trial. Trials. 2017 Feb 6;18(1):59. doi: 10.1186/s13063-017-1802-1. PMID 28166828